CLINICAL TRIAL: NCT02041975
Title: Investigating the Effects of Prebiotic-based Snacks on Perceived Feelings of 'Satisfaction' and on the Balance of Bacteria in the Human Gut (NutriSAT)
Brief Title: Effects of Prebiotic-based Snacks on the Gut Microbiota and Perceived 'Satisfaction'
Acronym: NutriSAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Roquette Freres (Industry)
Responsible Party: Principal Investigator, Mark Hobden, Mr, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H5117800; Ethics No. 11/08 (Other: University of Reading)
Record Dates: First submitted 2014-01-10; First posted 2014-01-22 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Obesity
Keywords: Prebiotics; Gut health; Satisfaction
MeSH Terms: conditions — Obesity; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prebiotic (Experimental): Nutriose FB06 14g/day
  Interventions: Dietary Supplement: Nutriose FB06
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutriose FB06 — Wheat dextrin soluble fibre
  Arms: Prebiotic
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
To determine the effects of prebiotic 'snacks' on gut health and satisfaction between meals

DETAILED DESCRIPTION:
The role of the bacteria that reside in the human gut play in human health and disease is of increasing importance. Evidence gathered over recent decades' shows that certain bacteria can improve resistance to gut infections, reduce cholesterol levels, synthesise vitamins and improve the immune response. The potential to modulate the relative balance of these so-called 'beneficial' bacteria has been demonstrated through the use of certain fibre sources termed prebiotics. In addition there is interest to understand how snacks containing these fibre sources may affect levels of 'satisfaction' between meals. The current study will address these issues and lead to a greater understanding of the role that prebiotics may play in gut health and overall metabolism.

ELIGIBILITY:
Inclusion Criteria -

* Aged between 22 and 55 years
* Healthy (no medical conditions in the last 12 months)
* BMI between 22.0 and 27.9 kg/m2
* Non-smokers
* Not a vegetarian or vegan
* No antibiotics in the last 6 months
* Not donated more than 350 ml blood in 4 months prior to or following study

Exclusion Criteria -

* Had surgery or suffered a medical condition affecting the circulatory, nervous or digestive systems in the previous 12 months
* Had suffered a myocardial infarction or stroke in the previous 12 months
* Suffer from any blood-clotting disorder or prescription of any medication affecting blood clotting
* Suffer from any metabolic disorders (e.g. diabetes, metabolic syndrome or hypertension)
* Any requirement to take long-term medication, especially those active on the gastro-intestinal tract or for cardio-vascular disease [including proton pump inhibitors (e.g. Omeprazole, Esomeprazole, Lansoprazole or Pantoprazole), non-steroidal anti-inflammatory drugs (e.g. acetylsalicylic acid, ibuprofen or diclofenac) or anti-anxiety medication (e.g. benzodiazepine)]
* Use of antibiotics within the previous 6 months
* Any dietary restrictions or on a weight reducing diet
* Irregular eating patterns and those not consuming breakfast
* Any food allergies (e.g. milk protein allergies) or intolerances (e.g. lactose)
* Use of medication which affects food intake or behaviour (e.g. anti-depressants)
* Use of medication likely to affect taste, smell or appetite
* Use of cholesterol lowering drugs/functional foods (e.g. Flora pro-activ)
* Dietary fibre consumption > 20 g/d
* Those that dislike the study foods and beverages
* Three Factor Eating Questionnaire (TFEQ) Factor 1 score >13
* Use of any vitamin supplements or fish oil capsules
* A history of alcohol or drug misuse (the average daily number of units of alcohol considered as acceptable is 2-3 units women; 3-4 units men)
* Smoking
* Athletes in training (> 8 h exercise/week)
* Amount of sleep each night (<5 hours/night)
* Females who are breast-feeding, may be pregnant, or if of child-bearing potential and are not using effective contraceptive precautions
* Involvement in a study involving an experimental drug/medication within 4 weeks prior to entry to the study
* History of chronic constipation or diarrhoea, or other chronic gastrointestinal complaint (e.g. irritable bowel syndrome)
* Intake of other supplementary prebiotics (such as oligosaccharides, e.g. FOS, GOS) or probiotics, drugs active on gastrointestinal motility such as antidiarrheals (e.g. medicines containing loperamide, bismuth subsalicyte or atropine/diphenoxylate), medication for abdominal pain and intestinal discomfort (e.g. duspatalin) or laxatives of any class (medications containing e.g. polyethylene glycol 3350, bisacodyl, methylcellulose or lactulose) during or within the four weeks prior to the start of the study
* Aged below 22 or over 55 years
* Have a Body Mass Index (BMI) of less than 22 or more than 27.9 kg/m2 [for volunteers of Asian origin; BMI of less than 21, or between to 23 to 25, or above 27 kg/m2].
* Blood pressure > 160/90 mmHg
* Vegan or vegetarian
* Donated > 350 ml of blood within the 4 months prior to the study or plan on donating > 350 ml of blood within the 4 months following the study.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Differences in perceived appetite (assessed using visual analogue scales) | Within 18 months

SECONDARY OUTCOMES:
Alterations to the relative balance of bacterial groups in faeces (assessed using flow cytometry) | Within 18 months

OTHER OUTCOMES:
Changes to metabolite and gut hormones responses in plasma (measured using ELISA and other assays) | Within 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Orla Kennedy, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Hobden MR, Commane DM, Guerin-Deremaux L, Wils D, Thabuis C, Martin-Morales A, Wolfram S, Diaz A, Collins S, Morais I, Rowland IR, Gibson GR, Kennedy OB. Impact of dietary supplementation with resistant dextrin (NUTRIOSE(R)) on satiety, glycaemia, and related endpoints, in healthy adults. Eur J Nutr. 2021 Dec;60(8):4635-4643. doi: 10.1007/s00394-021-02618-9. Epub 2021 Jun 25. PMID 34170392